CLINICAL TRIAL: NCT05546151
Title: A Double-blind, Placebo-controlled, Randomized, Multiple Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of BMS-986322 in Healthy Participants of Japanese Descent
Brief Title: A Study to Assess the Safety and Tolerability of BMS-986322 in Healthy Participants of Japanese Descent
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM032-042
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Healthy Participants
Keywords: BMS-986322; Japanese descent

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort J1 (Experimental)
  Interventions: Drug: BMS-986322; Other: Placebo for BMS-986322
- Cohort J2 (Experimental)
  Interventions: Drug: BMS-986322; Other: Placebo for BMS-986322
- Cohort J3 (Experimental)
  Interventions: Drug: BMS-986322; Other: Placebo for BMS-986322

INTERVENTIONS:
Drug: BMS-986322 — Specified dose on specified days
Other: Placebo for BMS-986322 — Specified dose on specified days

SUMMARY:
The purpose of this study is to assess the safety and tolerability of multiple ascending oral doses of BMS-986322 in healthy participants of Japanese descent.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be of Japanese descent (both biological parents are ethnically Japanese).
* In the opinion of the investigator, is a healthy participant, without any clinically significant abnormalities in their medical history, physical examination, ECGs, or clinical laboratory assessments determinations.
* Women should be of non-childbearing potential.

Exclusion Criteria:

* Any significant acute or chronic medical illness.
* Current or recent (within 3 months of study drug administration) gastrointestinal disease that could impact upon the absorption of study drug.
* Any major surgery within 90 days of study drug administration.

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-04-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with serious adverse events (SAEs) | Up to 7 weeks
Number of participants with adverse events (AEs) leading to discontinuation | Up to 7 weeks
Number of deaths | Up to 7 weeks
Number of participants with AEs | Up to 7 weeks
Number of participants with electrocardiogram (ECG) abnormalities | Up to 7 weeks
Number of participants with vital sign abnormalities | Up to 7 weeks
Number of participants with physical examination abnormalities | Up to 7 weeks
Number of participants with clinical laboratory abnormalities | Up to 7 weeks

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Day 1 and Day 14
Time of maximum observed plasma concentration (Tmax) | Day 1 and Day 14
Area under the concentration-time curve within a dosing interval (AUC[TAU]) | Day 1 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Anaheim Clinical Trials Llc, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html.

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com